CLINICAL TRIAL: NCT05483062
Title: Effectiveness of Toothpaste Containing the Active Ingredient of Galla Chinensis Extract on Treating Dentin Hypersensitivity '' A Randomized Clinical Trial ''
Brief Title: Effectiveness of Toothpaste Containing the Active Ingredient of Galla Chinensis Extract on Treating Dentin Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ibram ibrahim morkous henein, principal investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Minia University Dentistry
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Tooth Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Galla chinensis; Tin Fluorides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- toothpaste with active ingredient of galla chinensis (Experimental)
  Interventions: Other: galla chinensis
- toothpaste with stannous fluoride (Active Comparator)
  Interventions: Other: Stannous fluoride

INTERVENTIONS:
Other: galla chinensis — toothpaste
  Arms: toothpaste with active ingredient of galla chinensis
Other: Stannous fluoride — Toothpaste
  Arms: toothpaste with stannous fluoride

SUMMARY:
This clinical trial was conducted to compare the desensitizing effect of toothpaste containing the active ingredient of an extract of Galla chinensis and toothpaste containing fluoride in patients with dentin hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Overall good oral hygiene status.
* Participants show tooth neck abrasion or gingival retraction.
* Patients have subjective dentin hypersensitivity (at least 1 tooth) after using airflow.
* No history of periodontal treatment, including periodontal surgery, in the past year.
* Written informed consent

Exclusion Criteria:

* Patient with severe periodontitis or severe erosion damage.
* Patients with a compromised medical history, or had received therapeutic irradiation to the head and neck region.
* Medically compromised patients where pain levels would be compromised.
* If analgesics or antibiotics have been administrated by the patient during the past 12 hours preoperatively as it might alter their pain perception.
* Patients reporting bruxism or clenching in order to avoid further pressure on an already hypersensitive tooth inducing subsequent irritation and inflammation.
* Teeth that show association with acute periapical abscess and swelling.
* Greater than grade I mobility or pocket depth greater than 5mm.
* Non-restorable teeth or hopeless teeth.
* Immature teeth.
* Radiographic evidence of external or internal root resorption.
* Alcoholic and smoker patients.
* Pregnant or breastfeeding ladies.
* Patients having physical disabilities, or who are unable to brush their teeth
* Patients who have a history of allergies to any personal oral care product or ingredient, or who are taking anti-inflammatory drugs within the previous month.
* Individuals who had sensitive teeth but with one of the following conditions will be excluded from the study, teeth with large restorations, abutment of teeth of removable partial dentures, dental caries, enamel cracks, leakage of fillings or other restorations, cracked 23
* teeth, dental pulp lesions, dental abscesses, pulpitis, and atypical facial pain.
* Patients had participated in a clinical trial within 6 months before commencement of this trial.
* Patients unable to return for recall appointment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Change of pain level in response to stimuli | 6 months follow up
  Teeth were evaluated at baseline (T0), 1week (T1), 2 weeks (T2), 4 weeks (T3), 3 months (T4), and 6 months (T5) after using different types of toothpastes using Visual Analog Scale (VAS) scoring from 0-10 while 0 mean no pain and 10 severe pain by sensitivity tests (schiff test )

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes